CLINICAL TRIAL: NCT06344260
Title: Neural Stem Cell Treatment for Amyotrophic Lateral Sclerosis: A Multicenter, Randomized Placebo Controlled and Biological Endpoints Clinical Trial
Brief Title: Neural Stem Cell Treatment for Amyotrophic Lateral Sclerosis (STEMALS)
Acronym: STEMALS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Casa Sollievo della Sofferenza IRCCS (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: hNSCALSII
Record Dates: First submitted 2024-03-18; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Neural Stem Cells; ALS; Biomarkers; ICV Surgery
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This is an approximate 24-months triple-blinded, randomized, controlled vs placebo, in three arms study (PHASE B). A preliminary 3+3 dose-escalation open-label phase (PHASE A) will be performed in order to test the toxicity of the two proposed cell doses.
  In the phase B three arms will be: 1) hNSCs 20 milion cells 2) hNSCs 40 milion cells 3) Saline (comparator)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In order to blind also the statistician that will analyse the results the protocol has been designed as a triple-blinded protocol. This means that both the researchers, which include neurologist, neurosurgeon and biologist, as well as the patients and the statisticians are unaware of whether the participant received the treatment or the placebo (only IMP Manufacturer QP is unblinded since release the cell drug to the use in the surgery room)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- hNSC 20*10^6 (Experimental): Inoculation of 20*10^6 neural stem cells into the right lateral ventricle through a silicone catheter
  Interventions: Procedure: human Neural Stem Cells (hNSC)
- hNSC 40*10^6 (Experimental): Inoculation of 40*10^6 neural stem cells into the right lateral ventricle through a silicone catheter
  Interventions: Procedure: human Neural Stem Cells (hNSC)
- Saline Solution (placebo) (Placebo Comparator): Inoculation of saline (placebo) into the right lateral ventricle through a silicone catheter
  The reservoir will be placed to all recruited patients in a first surgical session, after randomization half of the subjects will receive the drug product (further randomized for doses) and half the placebo. After three months (period of time considered the minimum for a correct clinical evaluation that does not risk having to exclude patients treated with placebo from subsequent treatment with cells due to excessive physical decline), patients that already received cells will also be infused with placebo while the others will be randomized and transplanted with one of the two cell doses previously mentioned
  Interventions: Procedure: Saline (Placebo)

INTERVENTIONS:
Procedure: human Neural Stem Cells (hNSC) — The patient is placed on a regular operating room table with or without rigid head fixation. Procedure will be performed whether under general anesthesia or sedation and local anesthesia. Image guidance will be registered using the frameless stereotactic AxiEM system. Image guidance will be used to perform ventricular cannulation with the catheter passed over an electromagnetic-tipped stylet, which is recognized and tracked by the navigation system. The correct placement of the catheter is verified by the egress of CSF. Finally the electromagnetic stylet will be removed and a Rickam reservoir connect to ventricular catheter. Operative time will be about 30 minute. A post-operative CT scan will be obtained in all patients to confirm the catheter position.
  Other Names: Injection of human neural stem cells into brain lateral ventricle
  Arms: hNSC 20*10^6; hNSC 40*10^6
Procedure: Saline (Placebo) — The patient is placed on a regular operating room table with or without rigid head fixation. Procedure will be performed whether under general anesthesia or sedation and local anesthesia. Image guidance will be registered using the frameless stereotactic AxiEM system. Image guidance will be used to perform ventricular cannulation with the catheter passed over an electromagnetic-tipped stylet, which is recognized and tracked by the navigation system. The correct placement of the catheter is verified by the egress of CSF. Finally the electromagnetic stylet will be removed and a Rickam reservoir connect to ventricular catheter. Operative time will be about 30 minute. A post-operative CT scan will be obtained in all patients to confirm the catheter position.
  Other Names: Injection of saline into brain lateral ventricle
  Arms: Saline Solution (placebo)

SUMMARY:
A Not for Profit Phase II Study to Evaluate Safety, Efficacy and Biomarkers secondary endpoints of Human Neural Stem cell intracerebroventricular transplantation in amyotrophic lateral sclerosis patients: a randomized, placebo controlled, triple blind study.

This is an approximate 24-months study (PHASE B) consisting, per patient, of a 30-day screening period, 12-month enrollment and follow up period. A preliminary 3+3 dose-escalation open-label phase (PHASE A) will be performed in order to test the toxicity of the two proposed cell doses. The study will be stopped when all the subjects included in the treatment period complete the study visits. The study uses an ATMP, for that reason all the patients follow up will be prosecuted long life.

DETAILED DESCRIPTION:
Phase A: Open, monocentric safety, dose-finding study: The hNSCs will be produced by the UPTA (Unità Produttiva per Terapie Avanzate) of "Casa Sollievo della Sofferenza" according to GMP guidelines and injected using an Ommaya reservoir which will be removed immediately after the transplant procedure. The reservoir consists of an indwelling ventricular catheter with a dome-shaped collapsible silicone reservoir port positioned under the scalp. The distal end of the catheter is surgically positioned into the ipsilateral ventricle and connected to the reservoir. Six patients affected by ALS will be consecutively enrolled after pre- and screening visits. Thereafter, the first three patients will receive 20 million of hNSCs. If none of the three patients will present a serious adverse event classified as related to the study treatment, the dose level will be escalated up to 40 million of hNSCs for the next and last cohort of three patients. An Independent Data Safety Monitoring Board (DSMB) will oversee the safety of the Study Subjects on an ongoing basis, will review all safety data and issue a final recommendation at the end of this phase. Phase B: randomized, controlled vs placebo, in three arms, with two different doses of 20 and 40 *10^6 cells transplanted using an Ommaya reservoir. The reservoir will be placed to all recruited patients in a first surgical session, after randomization half of the subjects will receive the drug product (further randomized for doses) and half the placebo. After three months, patients that already received cells will also be infused with placebo while the others will be randomized and transplanted with one of the two cell doses previously mentioned. This secondary randomization will be performed to provide experimental treatment to all patients and is not intended as a second stage of a cross-over study. In the second surgical session the Ommaya reservoir will be removed and patients will be monitored for 3 months after that.

ELIGIBILITY:
Inclusion Criteria:

1. Patient provides written informed consent, informed consent signature collection prior to any study procedure (patient has good acceptance and understanding of the informed consent);
2. Definite, probable diagnosis according to the revised El Escorial criteria;
3. Age: 18-65 years;
4. FVC >70%;
5. Onset ≤ 24 months;
6. Patients with an ALSFRS-R score of at least 26; overall, including a score of at least 2 on each of the 1-9 ALSFRS-R individual component items and of at least 3 of the 10-12 individual components items;
7. Evidence of fast progression of the disease. We exclude slow progressors at the time of screening defined as Patient with an ALSFRS-R total score progression between onset of the disease and screening of < 0.3 per month. We document the fast progression of the disease defined as ALSFRS-R total score decrease of ≥ 1 point per month during a 12 week run-in period between screening and randomization;
8. Patient should be on a stable dose of Riluzole for > 30 days from pre-screening visit or not taking riluzole at all, nor plan to begin riluzole during the study period;
9. Patient is medically able to tolerate transient immunosuppression regimen;
10. Presence of a willing and able caregiver who understands the need to attend all follow-up visits, even if mobility declines.

Exclusion Criteria:

1. Psychiatric disease or other neurological diseases different from ALS;
2. Evidence of any concurrent illness or treatments limiting the safety to participate or any condition that the neurosurgeon feels may pose complications for the surgery;
3. Cancer within the previous 10 years;
4. Immunosuppressive therapy within 12 weeks of screening; active autoimmune disease or infection (including hepatitis B, hepatitis C, or HIV);
5. Cognitive impairment;
6. Contraindications to perform MRI scans, CSF withdrawal and Skin biopsy;
7. Patient unable to understand informed consent form;
8. Pregnancy and breast feeding;
9. Patient has been treated previously with any stem cell or somatic cells therapy;
10. Patient has participated in another clinical treatment trial or received other experimental medications outside of a clinical trial within 1 month prior to start of this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Safety of treatment | From date of enrollment until 12 month.
  safety assessed with respect to the incidence of treatment-emergent AEs (TEAEs) and serious AEs (SAEs) over the whole study period

SECONDARY OUTCOMES:
Biological Endpoints | Samples for biological endpoints will be taken at treatment, 1, 3, and 6 months after treatment
  To evaluate the biological activity of hNSC treatment by measuring the levels of selected pharmacodynamics biomarkers in CSF and serum. Data will be statistically assessed for significance by either Student t test or analysis of variance as applicable. A p value of less than 0.05 will be considered statistically significant. Candidate markers include: lNf, GFAP, NF1, VEGF, Osteopontin, CXCL13, Cystatina, MCP-1 BDNF, YKL-40, IL-6, TNF-a, IL-17, TDP43 TAU In parallel to the clinical evaluation of hNSCs efficacy we will also develop patient-specific cell models in order to individuate molecular and cellular mechanisms supporting the putative therapeutic action of hNSCs treatment. These models will be derived from blood or skin cells of the patients recruited in the trial in order to produce iPS cells, then differentiated in NSCs.
  disease

CONTACTS AND LOCATIONS:
Overall Officials: Angelo L Vescovi, PhD, Study Director — Scientific Director Fondazione IRCCS "Casa Sollievo della Sofferenza"
Locations (4):
- Italy (4):
  - Casa Sollievo Della Sofferenza IRCCS, San Giovanni Rotondo, Foggia
  - Centro SLA Azienda Ospedaliera Università Maggiore della Carità, Novara
  - Azienda Ospedaliera di Padova, Padua
  - Azienza Ospedaliera Universitaria - Policlinico "P. Giaccone" Università degli Studi di Palermo, Palermo

IPD SHARING:
Plan to Share IPD: No